CLINICAL TRIAL: NCT00368225
Title: Transplant-Related Accelerated Progression of Hepatitis C (TRAP-C)
Brief Title: Transplant-Related Accelerated Progression of Hepatitis C
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060193; 06-CC-0193
Record Dates: First submitted 2006-08-23; First posted 2006-08-24 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-01-22

CONDITIONS: Hepatitis C; Cirrhosis
Keywords: Viral Hepatitis; Hepatitis C; HCV; Liver Transplant; Renal Transplant; Kidney Transplant
MeSH Terms: conditions — Hepatitis C; Fibrosis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will explore why severe scarring of the liver (cirrhosis) develops so rapidly in hepatitis C-infected patients who have had a liver transplant and possibly in kidney transplant patients as well. The hepatitis C virus (HCV) can cause cirrhosis in about 20 percent of infected persons. Generally, it takes 20 years or more for cirrhosis to develop. After liver transplantation, however, patients may develop cirrhosis in as little as 5 years. Cirrhosis does not develop as rapidly in kidney transplant patients, but it may develop faster than in people who do not undergo transplantation. The study will look at the possible role of immune-suppressing medications given to liver and kidney transplant patients in increasing the severity of hepatitis C infection and in speeding the cirrhotic process.

Patients 18 years of age and older with chronic HCV infection who require a liver transplant for end-stage liver disease or a kidney transplant for kidney failure may be eligible for this study. Liver transplant patients are recruited from the Inova Fairfax Liver Transplant Center in Fairfax, Virginia, and from the Georgetown University Medical Center Liver Transplant Institute in Washington, D.C. Kidney transplant patients are recruited from the Transplantation Branch of the National Institute of Diabetes and Digestive and Kidney Diseases.

Participants undergo the following procedures:

* Regular care: As part of their regular transplant-related treatment, patients have a medical history, physical examinations and blood draws before their transplant and on regularly scheduled visits after the transplant.
* Blood draws for research: Special blood tests are done to measure the immune response to HCV. They measure the amount of HCV in the blood, the number of HCV strains present and how they change over time and the HCV antibodies in the blood.
* Liver biopsies: This procedure is done at 3 months, 1 year, 3 years and 5 years after the transplant to determine the extent of scarring of the liver and to study the immune responses within the liver, the proportion of liver cells infected with HCV and the presence of scar-producing cells. The biopsy is done during a 1- to 2-day inpatient hospital stay. The patients are given a sedative medication through a vein before the procedure. The skin over the biopsy site is numbed and the biopsy needle is passed rapidly into and out of the liver to collect a small sample of liver tissue for study.
* Apheresis: This procedure is done to collect a large number of white blood cells needed to test the immune response to the HCV. On the day before each liver biopsy, blood is drawn through a needle from a vein in one arm and run through a machine that separates and collects the white cells. The red cells and plasma are returned to the patient's body through the same needle or a second needle in the other arm.

DETAILED DESCRIPTION:
Nearly all patients with hepatitis C virus (HCV) related end-stage liver disease who receive an orthotopic liver transplant (OLT) develop hepatitis C reinfection of the graft after transplantation. Most of these patients will progress to chronic hepatitis and 20-30% will experience a rapid progression to cirrhosis. It is unclear why it generally takes 20 or more years for progression to cirrhosis after the initial HCV infection, but as little as five years after OLT. Additionally, it is paradoxical that hepatitis C, which is thought to be immune-mediated, should advance more rapidly in patients who are immune suppressed. Rapid fibrosis progression post-transplantation is likely related to complex interactions between viral factors, host immune responses and induction and maintenance of immunosuppression for the prevention of graft rejection.

This study has been designed as an observational, hypothesis-generating pilot study of patients with chronic hepatitis C requiring organ transplantation and concomitant immunosuppression. Patients who require a liver-transplant for chronic hepatitis C-related end-stage liver disease and patients with hepatitis C who require a kidney transplant for renal failure will be enrolled and followed for up to five years. Virologic, immunologic and intrahepatic parameters will be correlated with the level of immunosuppression, degree of fibrosis, progression to cirrhosis and liver-related deaths in study subjects. The objectives of this study are to: 1) determine the proportion of patients with hepatitis C that progress to bridging fibrosis or cirrhosis at three and five years after liver or kidney transplantation (rapid-progressors); 2) compare virologic, host-immune and intrahepatic factors in rapid-progressors to non-progressors and slow progressors; 3) characterize the relationship between general and HCV-specific immune responses and the extent of liver fibrosis; and 4) develop a predictive model that discriminates between rapid-progressors and non- or slow-progressors.

ELIGIBILITY:
* INCLUSION CRITERIA

To fulfill criteria for study entry, the patient must:

* be 18 years of age or older.
* have detectable HCV RNA
* require orthotopic liver transplantation for chronic hepatitis C induced cirrhosis or require renal transplantation for end-stage kidney disease
* have a MELD score greater than 18 (for liver transplant patients) or have an otherwise high probability of receiving a liver or kidney transplant within six months of enrollment based on assessment by the clinical transplant team at each hospital.
* be able/willing to travel to the collaborating center for blood sampling prior to liver or kidney transplantation, and at 2, 3, 4, 5, 6, 8, 12, 16, 24 weeks after transplantation and then bi-annually until the end of the study at 5 years
* be willing to have study-related liver biopsies at 3 months, and then 1, 3 and 5 years after transplantation
* provide informed consent.

EXCLUSION CRITERIA:

To fulfill criteria for study entry, the patient must NOT:

* be HIV or Hepatitis B virus (HBsAg) positive
* receive a liver graft from an anti-HCV antibody positive or HBV core positive donor
* have other forms of liver disease including primary biliary cirrhosis, autoimmune hepatitis, hemochromatosis and Wilson's Disease
* have hepatocellular carcinoma if any single lesion is 5 cm. or more or if there are 3 or more lesions exceeding 3 cm.
* be on immunomodulatory medications such as corticosteroids within four weeks of collection of blood for pre-transplant baseline laboratory testing
* have been diagnosed with any hereditary or acquired immunodeficiency state prior to liver or kidney transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-06-22; Study Completion 2009-01-22

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Georgetown University, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Inova Fairfax Hospital, Falls Church, Virginia

REFERENCES:
- [Background] Alter MJ, Kruszon-Moran D, Nainan OV, McQuillan GM, Gao F, Moyer LA, Kaslow RA, Margolis HS. The prevalence of hepatitis C virus infection in the United States, 1988 through 1994. N Engl J Med. 1999 Aug 19;341(8):556-62. doi: 10.1056/NEJM199908193410802. PMID 10451460
- [Background] Davis GL. Chronic hepatitis C and liver transplantation. Rev Gastroenterol Disord. 2004 Winter;4(1):7-17. PMID 15029106
- [Background] Sheiner PA, Schluger LK, Emre S, Thung SN, Lau JY, Guy SR, Schwartz ME, Miller CM. Retransplantation for recurrent hepatitis C. Liver Transpl Surg. 1997 Mar;3(2):130-6. doi: 10.1002/lt.500030205. PMID 9346726